CLINICAL TRIAL: NCT04371159
Title: A Comparative, Controlled Study to Evaluate the Clinical Accuracy of the Velieve U.S. UTI Urine Analysis Test System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-Velieve-MC-02
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Velieve U.S. (Experimental): Each participant will test their urine sample using the Velieve U.S. device
  Interventions: Device: Velieve U.S.

INTERVENTIONS:
Device: Velieve U.S. — The Velieve U.S. is a home use, in-vitro diagnostic (IVD) device. The device is used for the semi-quantitative detection of blood and leukocytes, and the qualitative detection of nitrites in urine.

SUMMARY:
The Velieve U.S. UTI Urine Analysis Test System (henceforth Velieve U.S.) is composed of a kit and a smartphone application. The device will be provided to the subject in a simulated home-use environment. All subjects will be asked to complete the urine test by following the application guidance,including providing a urine sample and scanning the urine strip after placing it on the Color-Board. The user will also complete a questionnaire to collect information regarding the use of the Velieve U.S. device. Following the usability test performed by the lay user, the subject's urine sample will be tested by the professional user using the comparator device.

The use of the Velieve U.S. device will be evaluated for identified risks. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-80 years of age;
* Subjects who are healthy or:
* Subjects with a medical condition that normally present with an abnormal concentration of Leukocytes, Nitrites and Blood: (examples of such conditions include the following):

  * Urinary tract infection (UTI)
  * Patients with suspected or known occult blood in urine
  * Pregnant women
  * Other relevant conditions
* Subjects with any pathological findings which might be identified by the urine test (according to the physician discretion)
* Subject is capable and willing to provide informed consent;
* Subject has facility with both hands;
* Subject is capable and willing to adhere to the study procedures.
* Subject is familiar with the use of a smartphone
* Subject is capable of comprehending and following instructions in English

Exclusion Criteria:

* Subject has dementia.
* Subject has mental disorders.
* Subject cannot collect urine in a receptacle.
* Subject is visually impaired (cannot read the user manual).
* Any additional reason the study physician believes disqualifies the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the % agreement of the Velieve U.S., tested by the lay user, as compared to a comparator device, tested by a professional user. | 11 months

SECONDARY OUTCOMES:
Evaluation of the Velieve U.S. usability success rate, by potential lay users under actual use conditions. | 11 months

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Trials, LLC, West Palm Beach, Florida, United States